CLINICAL TRIAL: NCT01593787
Title: A Multi-center, Open Label Study for Evaluation of the Safety, Tolerability and Efficacy of 8-week Treatment With LCZ696 in Japanese Hypertensive Patients With Renal Dysfunction
Brief Title: Safety and Tolerability and Efficacy of LCZ696 in Japanese Hypertensive Patients With Renal Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696A1304
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension With Renal Dysfunction
Keywords: Hypertension; Renal dysfunction; LCZ696
MeSH Terms: conditions — Hypertension; Renal Insufficiency | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LCZ696 100 mg (Experimental): All participants were started on LCZ696 100 mg once daily on day 1.
  Interventions: Drug: LCZ696
- LCZ696 200 mg (Experimental): All participants were started on LCZ696 100 mg once daily on day 1. For participants who did not achieve msDBP <80 mmHg and msSBP <130 mmHg at or after week 2 and had no signs of safety concerns at specified visits during the treatment epoch, the LCZ696 dose was increased to LCZ696 200 mg.
  Interventions: Drug: LCZ696
- LCZ696 400 mg (Experimental): All participants were started on LCZ696 100 mg once daily on day 1. For participants who received LCZ696 200 mg and did not achieve msDBP <80 mmHg and msSBP <130 mmHg at or after week 4 and had no signs of safety concerns at specified visits during the treatment epoch, the LCZ696 dose was increased to LCZ696 400 mg.
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696 — 100 mg, 200 mg, 400 mg tablets.

SUMMARY:
This study assessed the safety, tolerability, and efficacy of LCZ696 in hypertensive patients with renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Renal findings: Hypertensive patients with renal dysfunction and stable renal condition at least 4 weeks before screening visit.
* Satisfy office msSBP ≥140 mmHg and <180 mmHg at baseline.

Exclusion Criteria:

* Patients show msDBP ≥110 mmHg and/or msSBP ≥180 mmHg.
* History of angioedema, drug-related or otherwise, as reported by the patient.
* Any other following renal disorder:
* Patients show eGFR < 15mL/min/1.73m^2
* Patients on dialysis
* Patients who previously entered a LCZ696 study and had been randomized or enrolled into the active drug treatment epoch.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Japan (11):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Aira, Kagoshima-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Fujimino, Saitama
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo

REFERENCES:
- [Background] Ito S, Satoh M, Tamaki Y, Gotou H, Charney A, Okino N, Akahori M, Zhang J. Safety and efficacy of LCZ696, a first-in-class angiotensin receptor neprilysin inhibitor, in Japanese patients with hypertension and renal dysfunction. Hypertens Res. 2015 Apr;38(4):269-75. doi: 10.1038/hr.2015.1. Epub 2015 Feb 19. PMID 25693859

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg
Started | 6 | 8 | 18
Completed | 5 | 8 | 18
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total
Number analyzed (Participants) | 6 | 8 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (5.10) | 71.3 (8.80) | 62.3 (9.04) | 65.8 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 8
  Male | 4 | 4 | 16 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reported Adverse Events (Total Adverse Events, Serious Adverse Events and Death)
Description: Percentage of patients with total adverse events, serious adverse events and death were reported.
Time Frame: 8 weeks
Population: Safety Set: This set included all participants who received at least one dose of LCZ696. AE analysis was determined by actual treatment, i.e. the LCZ696 dose on the day in which the corresponding summary was targeting. Other safety analysis was determined by the maximum treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Total LCZ696: All participants who received LCZ696
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 32 | 26 | 18 | 32
Percentage of participants
  Adverse events (serious and non-serious) | 31.3 | 0 | 27.8 | 43.8
  Serious Adverse Events | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) at Week 8
Description: Sitting BP measurements were performed at screening through the end of study at every visit. Four separate sitting BP were obtained with a full two-minute interval between measurements.
Time Frame: baseline, 8 weeks
Population: Full Analysis Set (FAS): This set included all participants who entered the treatment epoch. Patients who were not qualified to enter the treatment epoch were excluded from the FAS provided those participants did not receive LCZ696.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 6 | 8 | 18 | 32
mmHg | -19.71 (12.314) | -27.19 (10.557) | -17.79 (10.701) | -20.50 (11.329)

3. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) at Week 8
Time Frame: baseline, 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 6 | 8 | 18 | 32
mmHg | -7.17 (4.690) | -9.94 (7.557) | -7.99 (6.385) | -8.32 (6.308)

4. Secondary Outcome: Percentage of Participants Achieving a Successful BP Control at Week 8
Description: A successful BP control was defined as msSBP <130 mmHg and msDBP <80 mmHg
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of Participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 6 | 8 | 18 | 32
Percentage of Participants | 66.7 | 37.5 | 5.6 | 25.0

5. Secondary Outcome: Percentage of Participants Achieving SBP Control at Week 8
Description: SBP control was defined as msSBP <130 mmHg.
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 6 | 8 | 18 | 32
Percentage of participants | 66.7 | 50.0 | 44.4 | 50.0

6. Secondary Outcome: Percentage of Participants Achieving DBP Control at Week 8
Description: DBP control was defined as msDBP <80 mmHg.
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 6 | 8 | 18 | 32
Percentage of participants | 83.3 | 62.5 | 27.8 | 46.9

7. Secondary Outcome: Percentage of Participants Achieving a Successful Response Rate in msSBP at Week 8
Description: Successful response rate was defined as msSBP <130 mmHg or a reduction of ≥20 mmHg from baseline
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 6 | 8 | 18 | 32
Percentage of participants | 66.7 | 75.0 | 50.0 | 59.4

8. Secondary Outcome: Percentage of Participants Achieving a Successful Response Rate in msDBP at Week 8
Description: Successful response rate was defined as msDBP <80 mmHg or a reduction of ≥10 mmHg from baseline.
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Total LCZ696
Number analyzed (Participants) | 6 | 8 | 18 | 32
Percentage of participants | 83.3 | 87.5 | 61.1 | 71.9

ADVERSE EVENTS:
Groups:
- LCZ 100 mg: LCZ 100 mg
- LCZ 400 mg: LCZ 400 mg
- LCZ 200 mg: LCZ 200 mg
Arm/Group | LCZ 100 mg | LCZ 400 mg | Total LCZ696 | LCZ 200 mg
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/18 | 0/32 | 0/26
Other Adverse Events (participants affected / at risk) | 5/32 | 5/18 | 9/32 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ 100 mg (N=32) | LCZ 400 mg (N=18) | Total LCZ696 (N=32) | LCZ 200 mg (N=26)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1 | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 5 | 1 | 6 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.